CLINICAL TRIAL: NCT01070238
Title: Explorative, Pilot Study With Cross-over Design on the Metabolic Response of Orally Applied Slow Released Carbohydrates in Diabetes Type 2 Patients
Brief Title: Metabolic Response of Slow Released Carbohydrates in Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Numico Research (Unknown)
Responsible Party: Thomas Linn/Principal Investigator, University of Giessen
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: RA.4240.UKGiessen.021219.B
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2002-11

CONDITIONS: Type 2 Diabetes
Keywords: Isomaltulose; Slow Released Carbohydrates; Postprandial Glucose Metabolism; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — isomaltulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Isomaltulose

SUMMARY:
The study was conducted

1. to investigate the superiority of isomaltulose in reduction of postprandial hyperglycemia
2. to describe the kinetics of glucose absorption after a load of isomaltulose
3. to demonstrate the safety of a single load of isomaltulose compared to sucrose in type 2 diabetic patients.

DETAILED DESCRIPTION:
Epidemiological studies have shown that postprandial hyperglycemia is associated with atherosclerotic diseases. Therefore, therapeutic strategies to reduce postprandial hyperglycemia are desirable. An effective way to improve postprandial glucose level is the use of carbohydrates with low glycemic index. Isomaltulose is a reducing disaccharide occurring naturally in honey and sugar cane juice, including products derived thereof. It is an isomer of sucrose and composed of glucose and fructose linked alpha-1,6 instead of alpha-1,2.

Isomaltulose has been reported to be digested more slowly than sucrose. Due to this property, lower and slower increases in blood glucose responses are expected for isomaltulose than sucrose. Early studies have demonstrated attenuated glycemic and insulin responses after isomaltulose ingestion than after sucrose. This study was performed to describe the postprandial glucose metabolism more comprehensively after bolus administration of different doses of isomaltulose compared to sucrose in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: type 2 diabetes according to WHO/ADA criteria for more than 1 yr
* Adults aged 18-75 years old
* HbA1c < 8%, fasting blood glucose < 140 mg/dl
* For at least 2 months prior to visit 1, subjects must have been on a stable antidiabetic therapy regimen
* Subjects willing to perform home blood glucose monitoring and to otherwise comply with study protocol requirements

Exclusion Criteria:

* Type 1 diabetes mellitus
* Pregnant or lactating women or women planning to become pregnant
* Women who become pregnant will be withdrawn from the study
* Clinically significant heart, liver, lung, or kidney disease
* Drug or alcohol abuse
* Concomitant therapy with systemic glucocorticoids or acarbose
* Subjects unable to adhere to instructions during the qualification phase

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Lower postprandial glucose and insulin responses after isomaltulose ingestion than after sucrose

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Giessen and Marburg, Giessen, Hesse, Germany

REFERENCES:
- [Derived] Ang M, Linn T. Comparison of the effects of slowly and rapidly absorbed carbohydrates on postprandial glucose metabolism in type 2 diabetes mellitus patients: a randomized trial. Am J Clin Nutr. 2014 Oct;100(4):1059-68. doi: 10.3945/ajcn.113.076638. Epub 2014 Jul 16. PMID 25030779